CLINICAL TRIAL: NCT03276247
Title: Ethnic and Genetic Factors of Iron Status in Women of Reproductive Age
Brief Title: Iron Status in Women of Reproductive Age Reproductive Age
Status: Completed | Type: Observational
Sponsor: Victor Gordeuk (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor-Investigator, Victor Gordeuk, Professor of Medicine, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Other Study IDs: HEIRS-womenrepage
Record Dates: First submitted 2017-09-01; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Iron Metabolism Disorders
MeSH Terms: conditions — Iron Metabolism Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Asian American non-pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as Asian American and non-pregnant/non-breastfeeding.
  Interventions: Other: observation
- African American non-pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as African American and non-pregnant/non-breastfeeding.
  Interventions: Other: observation
- Hispanic American non-pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as Hispanic American and non-pregnant/non-breastfeeding.
  Interventions: Other: observation
- White non-pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as white and non-pregnant/non-breastfeeding.
  Interventions: Other: observation
- Asian American pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as Asian American and pregnant or breastfeeding.
  Interventions: Other: observation
- African American pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as African American and pregnant or breastfeeding.
  Interventions: Other: observation
- Hispanic American pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as Hispanic American and pregnant or breastfeeding.
  Interventions: Other: observation
- White pregnant: Women 25 to 44 years of age recruited in a primary care setting and self reported as White and pregnant or breastfeeding.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Analyzed iron status, HFE mutations and ethnicity for women in five primary care centers in the United States and Canada using de-identified data from the HEIRS study.

DETAILED DESCRIPTION:
HEIRS included a cross-sectional screening study of 101,168 patients, 25 years of age or older, in the primary care setting. Participants were recruited from four centers in the U.S .and one in Canada from February 2001 to February 2003. We will evaluate results for women aged 25-44 years of age who are self-reported as Asian, Black, Hispanic or White. The lower detection limit for the serum ferritin (SF) assay in the HEIRS study was 15 μg/L and therefore the definition of iron deficiency will be SF concentration ≤ 15 μg/L. Elevated SF concentrations, possibly indicative of elevated iron stores, will be classified by two definitions: 1) SF concentration > 300 μg/L and 2) SF >200 μg/L in combination with TSAT >45%. Proportions will be compared by Pearson's chi-square. Logistic regression models will be used to identify independent associations with measures of iron deficiency and elevated iron stores.

ELIGIBILITY:
Inclusion Criteria:

1. primary care women included in the HEIRS study with in the age range of this study
2. Self designation as Asian American, African American, Hispanic American or White.

Exclusion Criteria:

1. Age >44 years
2. Self-described ethnicity other in than inclusion criterion 2.

Ages: 25 Years to 44 Years | Sex: Female
Age Groups: Adult
Study Population: Primary care women included in the HEIRS study.
Sampling Method: Non-Probability Sample
Enrollment: 22042 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Elevated serum ferritin | One measurement was made at the time of recruitment and this is the measurement that will be analyzed.
  Serum ferritin >300 ug/L
Elevated serum ferritin and transferrin saturation | One measurement was made at the time of recruitment and this is the measurement that will be analyzed.
  Serum ferritin >200 ug/L and transferrin saturation >45%
Iron deficiency | One measurement was made at the time of recruitment and this is the measurement that will be analyzed.
  Serum ferritin <15ug/L

CONTACTS AND LOCATIONS:
Overall Officials: Victor R Gordeuk, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordeuk VR, Brannon PM. Ethnic and genetic factors of iron status in women of reproductive age. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1594S-1599S. doi: 10.3945/ajcn.117.155853. Epub 2017 Oct 25. PMID 29070555